CLINICAL TRIAL: NCT00382863
Title: Prospective Evaluation of Elastic Restraint to LESSen the Effects of Heart Failure (PEERLESS-HF) Trial
Acronym: PEERLESS-HF
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Resources unavailable to continue study follow-up.
Sponsor: Paracor Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure
Keywords: heart failure; cardiac support; Paracor; HeartNet; PEERLESS-HF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): HeartNet and Optimal Medical/Device Therapy (e.g., medications and cardiac resynchronisation therapy)
  Interventions: Device: HeartNet Ventricular Support System
- Control (Active Comparator): Optimal Medical/Device Therapy alone (e.g., medications and/or cardiac resynchronisation therapy) (Note: For the purpose of the PEERLESS-HF study, optimal medical therapy is defined as the use of angiotensin converting enzyme (ACE) inhibitors and Beta blockers in the highest tolerable doses for three months prior to study enrollment, and Optimal device therapy is defined as cardiac resynchronization therapy (CRT) or cardiac resynchronization therapy-defibrillator (CRT-D) for at least three months prior to study enrollment, when indicated.)
  Interventions: Drug: Optimal Medical/Device Therapy

INTERVENTIONS:
Device: HeartNet Ventricular Support System — The HeartNet Implant is placed on the epicardial surface of the heart surrounding both the left and right ventricles.
  Other Names: cardiac support
  Arms: Treatment
Drug: Optimal Medical/Device Therapy — Optimal Medical/Device Therapy - For the purpose of the PEERLESS-HF study, optimal medical therapy is defined as the use of ACE inhibitors and Beta blockers in the highest tolerable doses for three months prior to study enrollment, and Optimal device therapy is defined as CRT or CRT-D for at least three months prior to study enrollment, when indicated.
  Other Names: heart failure medications
  Arms: Control

SUMMARY:
The purpose of this study is to determine if patients in the HeartNet Ventricular Support System with optimal medical and device therapy arm (Treatment group) show statistically significant improvement compared to patients in the optimal medical and device therapy alone arm (Control group) after 6 months of follow-up.

DETAILED DESCRIPTION:
In the United States alone, more than five million people suffer from heart failure (CHF) and an estimated 400,000 to 700,000 new cases are diagnosed each year. Caused by a variety of cardiac conditions, systolic heart failire (HF) is the end-stage of heart disease where the heart is failing as a pump. Once diagnosed with the disease, less than 50% of the patients live for five years, and less than 25% survive for more than ten years. The number of deaths in the United States from this condition has more than doubled since 1979, averaging more than 250,000 annually.

Paracor Medical, Inc. has developed an elastic prosthetic wrap that is designed to apply a gentle mechanical support to the failing heart. The Implant is a compliant elastic structure that is designed to conform to the epicardial surface of the right and left ventricles. It supports the heart throughout the cardiac cycle and was designed to offload the ventricles and reduce wall stress.

The objective of this clinical trial is to evaluate the safety and efficacy of the HeartNet Ventricular Support System with optimal medical and device therapy (Treatment group) when compared to optimal medical and device therapy (i.e., medications, cardiac resynchronisation therapy, pacemaker) alone (Control group) as treatments for patients with heart failure.

Efficacy of the HeartNet Ventricular Support System in the Treatment group compared to the optimal medical and device therapy Control group will be evaluated based upon cardiopulmonary tests (Peak VO2), six (6) minute walk distance and quality of life assessment, as measured by the Minnesota Living with Heart Failure (MLWHF) questionnaire.

Safety of the HeartNet Ventricular Support System in the Treatment group compared to the Control group will be evaluated based on the all-cause mortality rate.

Paracor Medical intends to submit data obtained in this clinical trial to support a Pre-Market Approval Application to the United States Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic heart failure at enrollment (American College of Cardiology [ACC]/American Heart Association [AHA] Stage C) due to ischemic or nonischemic dilated cardiomyopathy
2. On stable, evidence-based medical and device therapy for heart failure for 3 months prior to randomization <a> Pharmacological Therapy (as appropriate) <i> angiotensin converting enzyme (ACE) inhibitors or angiotensin II receptor blockers (ARB) for patients with ACE inhibitor intolerance or nitrate/hydralazine at the investigators discretion <ii> beta blockers <iii> diuretics, aldosterone inhibitors <b> Ejection fraction < or = to 35% while maintained on optimal medical therapy <c> Cardiac Resynchronization Therapy (CRT), Cardiac Resynchronization Therapy-Defibrillator (CRT-D) <i> If implanted with a CRT or CRT-D, it must be implanted > or = to 3 months before randomization <ii> If currently eligible or anticipated eligibility with a CRT or CRT-D within 6 months, the patient should not be enrolled in the study

Specific Qualifying Characteristics

1. Six (6) minute walk of 150 - 450m
2. Peak VO2 for males: 10.0-20.0 ml/kg/min; Peak VO2 for females: 9.0-18.0 ml/kg/min
3. Left ventricular end diastolic diameter (LVEDD) <85mm and index <40mm/m2 (LVEDD/BSA)
4. Heart failure duration > or = to 6 months

Exclusion Criteria:

Patient History

1. Heart failure due to a reversible condition
2. Hypertrophic obstructive cardiomyopathy (HOCM)
3. Left ventricular assist device (LVAD), intra-aortic balloon pump (IABP) or intravenous inotropes are required or the patient has end stage heart failure despite maintenance on best medical therapy
4. Myxoma
5. Active infection, sepsis, endocarditis, myocarditis or pericarditis
6. Myocardial infarction, stroke, transient ischemic attack, cardiac or other major surgery, or implantable cardioverter defibrillator (ICD) or pacemaker implantation in the 3 months prior to entry
7. Positive pregnancy test for pre-menopausal female
8. Less than 18 years or > or = to 75 years old
9. Hemoglobin level less than 10 gm/dL or creatinine >2.5 mg/dL
10. Uncontrolled medical conditions that increase surgical risk
11. Co-morbid condition that in the investigator's opinion reduces life expectancy to less than 2 years

Surgical or Anatomical Considerations

1. Heart measurement too large or small for Implant sizes
2. Restrictive cardiomyopathy
3. Not a candidate for sternotomy or standard thoracotomy surgical approaches
4. Expected to have adhesions from previous surgical procedures
5. History of constrictive pericarditis
6. Previously placed coronary artery bypass grafts (CABG) or anticipated need for coronary artery bypass grafting
7. Not a candidate for cardiopulmonary bypass
8. Anatomical mitral valve regurgitation of 2+ or greater at the time of enrollment
9. Pulmonary function testing with the following results: Forced expiratory volume (FEV1) <1L or if FEV1 is between 1 and 3L, forced expiratory volume divided by forced vital capacity (FEV1/FVC) <60%
10. Cardiac or thoracic condition that might require operative correction. Cardiac transplantation is not included in this exclusion criterion.
11. Other elective surgical procedure at the time of the index hospitalization or within 30 days, whichever is longer

Other

1. Any other medical condition that, in the judgment of the investigator, makes the patient a poor candidate for this procedure
2. Currently enrolled or has participated in the last 30 days in another therapeutic or interventional clinical study
3. Unwilling/unable to comply with follow-up
4. Unwilling/unable to give signed informed consent

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2006-10; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T. Abraham, MD, Principal Investigator — Chief, Division of Cardiovascular Medicine, The Ohio State University
Locations (35):
- United States (29):
  - University of Alabama Birmingham, Birmingham, Alabama
  - USC Keck School of Medicine, Los Angeles, California
  - University of California, San Francisco, Medical Center, San Francisco, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Christiana Care Health System, Newark, Delaware
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Midwest Heart Foundation, Lombard, Illinois
  - St. Vincent Hospital and Health Services, Indianapolis, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - University of Maryland, Division of Cardiology, Baltimore, Maryland
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Wayne State University/ Oakwood Hospital, Detroit, Michigan
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - St. Paul Heart Clinic, Saint Paul, Minnesota
  - Mid America Heart Institute, Kansas City, Missouri
  - BryanLGH Heart Improvement Program, Lincoln, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - The Stern Cardiovascular Center, Germantown, Tennessee
  - Tennessee Cardiovascular Research Institute, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - Inova Heart & Vascular Institute/ Fairfax Hospital, Falls Church, Virginia
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - McGill University Hospital Centre, Montreal, Quebec

REFERENCES:
- [Derived] Abraham WT, Anand I, Aranda JM Jr, Boehmer J, Costanzo MR, DeMarco T, Holcomb R, Ivanhoe R, Kolber M, Rayburn B. Randomized controlled trial of ventricular elastic support therapy in the treatment of symptomatic heart failure: rationale and design. Am Heart J. 2012 Nov;164(5):638-45. doi: 10.1016/j.ahj.2012.07.015. Epub 2012 Oct 2. PMID 23137493
- [Derived] Keteyian SJ, Brawner CA, Ehrman JK, Ivanhoe R, Boehmer JP, Abraham WT; PEERLESS-HF Trial Investigators. Reproducibility of peak oxygen uptake and other cardiopulmonary exercise parameters: implications for clinical trials and clinical practice. Chest. 2010 Oct;138(4):950-5. doi: 10.1378/chest.09-2624. Epub 2010 Jun 3. PMID 20522572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 29 investigational sites in the US and 6 investigational sites in Canada, between November, 2006 to September, 2009
Pre-assignment Details: 3 subjects were considered Roll-in (not randomized) and received treatment. Data from these subjects are not included in the results. Seven (7) subjects were randomized to the Treatment group but were not treated due to suspension of the study. These subjects are excluded from the data.
Groups:
- Treatment: HeartNet and Optimal Medical/Device Therapy
- Control: Optimal Medical/Device Therapy alone
Period: Overall Study
Arm/Group | Treatment | Control
Started | 96 | 114
Completed | 81 | 78
Not Completed | 15 | 36
Not completed — Death | 9 | 9
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 5 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 96 | 114 | 210
Age Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.2) | 54.5 (10.8) | 54.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 35 | 63
  Male | 68 | 79 | 147
Race (NIH/OMB) [Number; unit: participants] — Self-reported race. Since the participants were allowed to select more than one race, the sum of races is greater than the number of participants in each group.
  participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 2 | 3 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 16 | 20 | 36
    White | 76 | 93 | 169
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 1
New York Heart Association (NYHA) Classification [Number; unit: participants]
  NYHA I: Pts w/cardiac disease, w/o activity limit | 3 | 4 | 7
  NYHA II; Pts w/cardiac disease, slight limits | 49 | 53 | 102
  NYHA III; Marked limit to physical activity | 43 | 57 | 100
  NYHA IV; inability to have activity w/o discomfort | 1 | 0 | 1
Heart Failure Etiology [Number; unit: participants]
  Non-ischemic | 62 | 80 | 142
  Ischemic | 34 | 34 | 68
  Unknown | 0 | 0 | 0
Duration of Heart Failure (time) [Mean (Standard Deviation); unit: years] | 7.7 (6.2) | 6.5 (5.0) | 7.1 (5.6)
Cardiac Medications [Number; unit: participants] — Baseline information for specific cardiac medications was requested. Since most participants were on more than one medication, the sum of medications are greater than the number of participants in each group.
  participants
    ACE Inhibitors | 72 | 86 | 158
    Antiogensin Receptor Blockers | 27 | 24 | 51
    Beta Blockers | 94 | 114 | 208
    Diuretics (other than Spironolactone) | 81 | 100 | 181
    Aldosterone Inhibitors | 53 | 76 | 129
    Digoxin | 45 | 53 | 98
Medical History and Co-Morbidities [Number; unit: participants] — Baseline information on specific co-morbities was requested. Since many participants had more than one co-morbidity, the sum of co-morbidities are greater than the number of participants in each group.
  participants
    Systemic Hypertension | 49 | 53 | 102
    Pulmonary Hypertension | 16 | 14 | 30
    Diabetes Mellitus | 30 | 42 | 72
    Chronic Obstructive Pulmonary Disease (COPD) | 8 | 13 | 21
    Sleep Apnea | 28 | 30 | 58
    Asthma | 11 | 11 | 22
    Coronary Artery Disease with Angioplasty/Stent | 31 | 30 | 61
    Stroke TIA/Other Thromboembolic Events | 12 | 9 | 21
    Peripheral Vascular Disease | 3 | 1 | 4
    Myocardial Infarction | 35 | 33 | 68
    Ventricular Tachycardia | 28 | 40 | 68
    Atrial Fibrillation | 22 | 28 | 50
    Biventricular Pacemaker | 3 | 3 | 6
    Biventricular ICD | 41 | 57 | 98
    Pacemaker alone | 0 | 1 | 1
    ICD alone | 42 | 45 | 87
    ICD with Bradycardia Pacing Capability | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Responder Analysis - Peak Oxygen Uptake (Peak VO2)
Description: A participant was considered a "responder" if cardiopulmonary exercise testing demonstrated an improvement in peak VO2 of at least 1.0 ml/kg/min at 6 months as compared to baseline.
Time Frame: Baseline to 6 months
Population: The population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 91
participants | 31 | 35
Statistical Analysis 1: Comparison: Treatment vs Control; Null hypothesis = proportion of subjects in treatment group who successfully achieved an improvement of at least 1.0 ml/kg/min at 6 months is less than or equal to the Control group. Subjects who withdrew for cardiac-related reasons were classified as non-responders; Test type: Superiority or Other; p = 0.502, Fisher Exact; One-sided

2. Primary Outcome: Responder Analysis - Six (6) Minute Walk (6MW) Distance
Description: A participant was considered a "responder" if 6MW distance at 6 months was at least 45 meters more than at baseline.
Time Frame: Baseline to 6 months
Population: The population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 87 | 99
participants | 33 | 25
Statistical Analysis 1: Comparison: Treatment vs Control; The null hypothesis = the proportion of subjects in the treatment group who successfully achieved an improvement of at least 45 m at 6 months from baseline is less than or equal to that of the Control group. Withdrawals due to cardiac reasons are counted as non-responders; Test type: Superiority or Other; p = 0.044, Fisher Exact; One-sided

3. Primary Outcome: Responder Analysis - Minnesota Living With Heart Failure (MLWHF) Quality of Life Overall Score
Description: A participant was considered a "responder" if the MLHF overall score had improved by at least 7 points at 6 months as compared to baseline. THE MLHF questionnaire evaluates the impact of heart failure (HF) on a subject's physical, emotional, social and mental aspects of quality of life. Each of 21 questions about how much HF impacts daily activities is scored from 0-no impact to 5-very much (overall score can range from 0 to 105). Improvement is indicated by a decrease in score.
Time Frame: baseline to 6 months
Population: The population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 93 | 101
participants | 53 | 50
Statistical Analysis 1: Comparison: Treatment vs Control; The null hypothesis = the proportion of treatment subjects who successfully achieved an improvement of at least 7 points at 6 months is equal to or less than that of the control group. Withdrawals due to cardiac reasons are counted as non-responders; Test type: Superiority or Other; p = 0.184, Fisher Exact; One-sided

4. Primary Outcome: Number of Participant Deaths
Description: Total number of participants who died within 12 months of enrollment into the trial.
Time Frame: 12 months
Population: The population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 114
participants | 4 | 5
Statistical Analysis 1: Comparison: Treatment vs Control; The null hypothesis = survival in the treatment group at 12 months is not equivalent to that of the Control group; Test type: Non-Inferiority or Equivalence — Estimated survival for the treatment group was 93%. Estimated survival for the control group was 91.5%. A non-inferiority margin of 7.5%. Final test alpha level of 0.04825; p = 0.012, Exact binomial test; One-sided

5. Secondary Outcome: Change in New York Heart Association (NYHA) Functional Class
Description: Change in NYHA functional class between baseline and 6 months. "Maintained" means the participant's functional class remained the same as baseline. "Improved" means the participant's functional class improved (became lower in number) by at least one class. "Worsened" means the participant's functional class deteriorated (became higher in number) by at least one class.
Time Frame: baseline to 6 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 91 | 103
participants
  Improved | 37 | 29
  Maintained | 45 | 59
  Worsened | 9 | 15
Statistical Analysis 1: Comparison: Treatment vs Control; Class change from baseline; Test type: Superiority or Other; p = 0.052, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Quality of Life as Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The KCCQ is a 23-item questionnaire that quantifies physical function, symptoms, social function, self-efficacy/knowledge and quality of life. Scores range from 0 to 100, where higher scores reflect better health status. For this outcome measure, the difference between each participant's baseline and 6-month KCCQ scores was calculated. The mean change for each treatment arm is presented.
Time Frame: baseline to 6 months
Population: Population is intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 91 | 99
score on a scale | 12.6 (18.2) | 3.4 (16.8)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

7. Secondary Outcome: Change in Left Ventricular Mass
Description: The difference between each participant's baseline and 6-month echocardiographic measure of left ventricular mass was calculated. The median change for each treatment arm is presented. A decrease in mass is associated with an improvement in the participant's structural heart failure.
Time Frame: baseline to 6 months
Population: Population is intent to treat.
Measure: Median (Full Range); unit: grams
Arm/Group | Treatment | Control
Number analyzed (Participants) | 72 | 94
grams | -19.0 [-119.0 to 81.0] | 7.0 [-254.0 to 109.0]
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.032, Wilcoxon (Mann-Whitney); Two-sided

8. Secondary Outcome: Responder Analysis - Peak Oxygen Uptake (Peak VO2)
Description: A participant was considered a "responder" if cardiopulmonary exercise testing demonstrated an improvement in peak VO2 of at least 1.0 ml/kg/min at 12 months as compared to baseline.
Time Frame: baseline to 12 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 61 | 69
participants | 19 | 21
Statistical Analysis 1: Comparison: Treatment vs Control; Improvement of at least 1.0 ml/kg/min from baseline; Test type: Superiority or Other; p = 0.540, Fisher Exact; One-sided

9. Secondary Outcome: Responder Analysis - Six (6) Minute Walk (6MW) Distance
Description: A participant was considered a "responder" if 6MW distance at 12 months was at least 45 meters more than at baseline.
Time Frame: baseline to 12 Months
Population: Population is intent to treat
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 90 | 98
participants | 33 | 25
Statistical Analysis 1: Comparison: Treatment vs Control; Improvement of at least 45 m from baseline; Test type: Superiority or Other; p = 0.067, Fisher Exact; One-sided

10. Secondary Outcome: Responder Analysis - Minnesota Living With Heart Failure (MLWHF) Quality of Life Overall Score
Description: A participant was considered a "responder" if the MLHF overall score had improved by at least 7 points at 12 months as compared to baseline. THE MLHF questionnaire evaluates the impact of heart failure (HF) on a subject's physical, emotional, social and mental aspects of quality of life. Each of 21 questions about how much HF impacts daily activities is scored from 0-no impact to 5-very much (overall score can range from 0 to 105). Improvement is indicated by a decrease in score.
Time Frame: baseline to 12 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 91 | 101
participants | 52 | 43
Statistical Analysis 1: Comparison: Treatment vs Control; Improvement of at least 7 points from baseline; Test type: Superiority or Other; p = 0.031, Fisher Exact; One-sided

11. Secondary Outcome: Heart Failure Hospitalization - Actuarial Analysis
Description: Kaplan-Meier actuarial analysis of heart failure hospitalization (as classified by an independent Clinical Events Committee) within the first 12 months after enrollment
Time Frame: 12 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 114
participants | 9 | 19
Statistical Analysis 1: Comparison: Treatment vs Control; Kaplan-Meier actuarial time-to-first-event analysis; Test type: Superiority or Other; p = 0.109, Log Rank

12. Secondary Outcome: Change in Left Ventricular End Diastolic Volume
Description: The difference between each participant's baseline and 6-month echocardiographic measure of left ventricular end diastolic volume was calculated. The median change for each treatment arm is presented. A decrease in volume is associated with an improvement in the participant's structural heart failure.
Time Frame: baseline to 6 months
Population: Population is intent to treat.
Measure: Median (Full Range); unit: milliliters
Arm/Group | Treatment | Control
Number analyzed (Participants) | 89 | 98
milliliters | -3.8 [-108.1 to 127.5] | 10.9 [-143.7 to 176.3]
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.031, Wilcoxon (Mann-Whitney); Two-sided

13. Secondary Outcome: Change in Left Ventricular End Systolic Volume
Description: The difference between each participant's baseline and 6-month echocardiographic measure of left ventricular end systolic volume was calculated. The median change for each treatment arm is presented. A decrease in volume indicates an improvement in the participant's structural heart failure.
Time Frame: baseline to 6 months
Population: Population is intent to treat.
Measure: Median (Full Range); unit: milliliters
Arm/Group | Treatment | Control
Number analyzed (Participants) | 89 | 98
milliliters | -7.0 [-100.5 to 125.0] | 2.75 [-134.2 to 150.5]
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.179, Wilcoxon (Mann-Whitney); Two-sided

14. Secondary Outcome: Change in Ejection Fraction
Description: The difference between each participant's baseline and 6-month echocardiographic measure of left ventricular ejection fraction was calculated. The median change for each treatment arm is presented.
Time Frame: baseline to 6 months
Population: Population is intent to treat.
Measure: Median (Full Range); unit: percent
Arm/Group | Treatment | Control
Number analyzed (Participants) | 89 | 98
percent | 0.0 [-11.0 to 16.0] | 1.9 [-18.0 to 21.0]
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.070, Wilcoxon (Mann-Whitney); Two-sided

15. Secondary Outcome: Change in Left Ventricular End Diastolic Diameter
Description: The difference between each participant's baseline and 6-month echocardiographic measure of left ventricular end diastolic diameter was calculated. The median change for each treatment arm is presented. A decrease in diameter indicates an improvement in the participant's structural heart failure.
Time Frame: baseline to 6 months
Population: Population is intent to treat.
Measure: Median (Full Range); unit: centimeters
Arm/Group | Treatment | Control
Number analyzed (Participants) | 86 | 99
centimeters | -0.15 [-1.2 to 1.7] | 0 [-1.3 to 1.9]
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.015, Wilcoxon (Mann-Whitney); Two-sided

16. Secondary Outcome: Change in Left Ventricular End Systolic Diameter
Description: The difference between each participant's baseline and 6-month echocardiographic measure of left ventricular end systolic diameter was calculated. The median change for each treatment arm is presented. A decrease in diameter indicates an improvement in the participant's structural heart failure.
Time Frame: baseline to 6 months
Population: Population is intent to treat.
Measure: Median (Full Range); unit: centimeters
Arm/Group | Treatment | Control
Number analyzed (Participants) | 85 | 95
centimeters | -0.1 [-1.2 to 2.1] | 0.1 [-1.8 to 1.9]
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.032, Wilcoxon (Mann-Whitney); Two-sided

17. Secondary Outcome: Technical Success (Number of Treatment Arm Participants Successfully Implanted)
Description: "Technical success" refers to the ability to successfully deliver a device onto the epicardial surface and leave the device in a satisfactory position. Participants who did not undergo an implant procedure were excluded from this analysis.
Time Frame: 1 day
Population: Population is as treated, treatment only.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 93 | 0
participants | 92 |

18. Secondary Outcome: Heart Failure Death
Description: Number of participants who died within 12 months of enrolling in the study and whose cause of death was classified, by an independent Clinical Events Committee, as heart failure
Time Frame: 12 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 114
participants | 1 | 3
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.627, Fisher Exact; Two-sided

19. Secondary Outcome: Heart Failure Death - Actuarial Analysis
Description: Kaplan-Meier actuarial time-to-event analysis of deaths classified, by an independent Clinical Events Committee, as due to heart failure
Time Frame: 12 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 114
participants | 1 | 3
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.386, Log Rank

20. Secondary Outcome: Heart Failure Hospitalization
Description: Number of participants who experienced a heart failure hospitaliz (as classified by an independent Clinical Events Committee) within the first 12 months after enrollment.
Time Frame: 12 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 114
participants | 9 | 19
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.154, Fisher Exact; Two-sided

21. Secondary Outcome: All-Cause Hospitalization
Description: Number of participants who experienced a hospitalization (for any cause) within the first 12 months after enrollment. Within the Treatment Arm, hospitalization for the implant procedure was not included in this analysis.
Time Frame: 12 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 114
participants | 38 | 45
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 1.000, Fisher Exact; Two-sided

22. Secondary Outcome: All-Cause Hospitalization - Actuarial Analysis
Description: Kaplan-Meier actuarial time-to-first-event analysis of all-cause hospitalizations
Time Frame: 12 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 114
participants | 38 | 45
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.939, Log Rank

23. Secondary Outcome: Participants Experiencing Serious Adverse Events
Description: Number of participants who experienced a serious adverse event (as classified by an independent Clinical Events Committee) within the first 12 months after enrollment
Time Frame: 12 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 114
participants | 57 | 47
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.012, Fisher Exact; Two-sided

24. Secondary Outcome: Serious Adverse Events - Actuarial Analysis
Description: Kaplan-Meier actuarial time-to-first-event analysis of serious adverse events
Time Frame: 12 months
Population: Population is intent to treat.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 114
participants | 57 | 47
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.001, Log Rank

25. Secondary Outcome: Days Alive Out of Hospital
Description: Median number of days participants were not hospitalized within the first 12 months after enrollment. Within the Treatment Arm, hospitalization for the implant procedure was not included in this analysis.
Time Frame: 12 months
Population: Population is intent to treat.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 96 | 114
days | 365 [45 to 365] | 365 [149 to 365]
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.772, Wilcoxon (Mann-Whitney); Two-sided

ADVERSE EVENTS:
Time Frame: Participants were followed up to 3.5 years
Description: Events adjudicated per Clinical Events Committee (CEC) Charter by independent CEC.
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 57/96 | 47/114
Other Adverse Events (participants affected / at risk) | 85/96 | 71/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=96) | Control (N=114)
Worsening Heart Failure (Cardiac disorders) | 15 (42) | 27 (46) — Non-perioperative
Non-Ischemic Atrial/Ventricular Dysrhythmia (Cardiac disorders) | 10 (14) | 11 (17) — Non-perioperative
Cardiac Procedure (Cardiac disorders) | 9 (9) | 11 (12) — Non-perioperative
Other Cardiac Hospitalization (Cardiac disorders) | 8 (8) | 10 (12) — Non-perioperative
Syncope (Cardiac disorders) | 2 (2) | 2 (2) — Non-perioperative
Myocardial Infarct (Cardiac disorders) | 0 (0) | 2 (2) — Non-perioperative
Coronary Insufficiency/Acute Coronary Syndrome/Unstable Angina (Cardiac disorders) | 2 (2) | 1 (1) — Non-perioperative
Peripheral Vascular Disease (Vascular disorders) | 2 (3) | 0 (0) — Non-perioperative
Pulmonary or Vascular Emboli (Vascular disorders) | 0 (0) | 2 (2) — Non-perioperative
Stroke (Vascular disorders) | 2 (2) | 1 (1) — Non-perioperative
Transient Ischemic Attack (Vascular disorders) | 0 (0) | 1 (2) — Non-perioperative
Non-cardiac vascular surgery (Vascular disorders) | 1 (1) | 0 (0) — Non-perioperative
Other Vascular Condition (nonspecific) (Vascular disorders) | 0 (0) | 1 (1) — Non-perioperative
Non-cardiac/Non-vascular (General disorders) | 22 (32) | 24 (36) — Non-perioperative
Arrythmias (Cardiac disorders) | 6 (7) | 0 (0) — Perioperative, treatment only
Pericardial Syndrome (Cardiac disorders) | 5 (5) | 0 (0) — Perioperative, treatment only
Hypotension (Cardiac disorders) | 5 (5) | 0 (0) — Perioperative, treatment only
Blood Loss (Cardiac disorders) | 4 (5) | 0 (0) — Perioperative, treatment only
Worsening Heart Failure (Cardiac disorders) | 4 (4) | 0 (0) — Perioperative, treatment only
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
LV Laceration (Cardiac disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Chest Pain Syndrome (Cardiac disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Renal Failure/Insufficiency (Renal and urinary disorders) | 2 (2) | 0 (0) — Perioperative, treatment only
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) — Perioperative, treatment only
Prolonged Ventilation (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) — Perioperative, treatment only
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Bacteremia/Sepsis (Infections and infestations) | 5 (5) | 0 (0) — Perioperative, treatment only
Pneumonia (Infections and infestations) | 2 (4) | 0 (0) — Perioperative, treatment only
Dehydration (General disorders) | 2 (2) | 0 (0) — Perioperative, treatment only
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Gastroesophageal Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Laryngeal Granuloma (General disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Ileus (General disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Alcohol Withdrawal (General disorders) | 1 (1) | 0 (0) — Perioperative, treatment only
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) — Perioperative, treatment only
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=96) | Control (N=114)
Cardiovascular (Cardiac disorders) | 63 (117) | 46 (68)
Respiratory/Pulmonary (Respiratory, thoracic and mediastinal disorders) | 32 (38) | 22 (31)
Gastrointestinal (Gastrointestinal disorders) | 7 (11) | 9 (11)
Neurology (Nervous system disorders) | 9 (10) | 3 (3)
Renal (Renal and urinary disorders) | 9 (9) | 5 (5)
Hematology (Blood and lymphatic system disorders) | 6 (7) | 3 (4)
Genital-urinary (Renal and urinary disorders) | 4 (7) | 3 (3)
General (General disorders) | 47 (97) | 35 (73)

LIMITATIONS AND CAVEATS:
An interim analysis indicated trial futility based on a primary endpoint. Enrollment was suspended in July, 2009. Study was terminated as of April, 2011 due to insufficient resources.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No